# **Exergaming Improves Executive Functions in**

# **Patients with Metabolic Syndrome**

Date of the document: May/27/2019

Shanshan Wu<sup>1</sup>, Eunah Jo<sup>2</sup>, Hongqing Ji<sup>1</sup>, Kyung-Hee Kim<sup>3</sup>, Jung-Jun Park<sup>1</sup>, Bo Hyun Kim<sup>4\*</sup>,
and Kyoung Im Cho<sup>2,\*</sup>

<sup>1</sup>Division of Sport Science, Pusan National University, Busan 46241, Korea

<sup>2</sup>Department of Internal Medicine, Kosin University College of Medicine, Busan 49267, Korea

<sup>3</sup>Department of Cardiology, Sejong General Hospital, Bucheon 22972, Korea

<sup>4</sup>Department of Internal Medicine, Pusan National University Hospital and Biomedical

14 Running Title: Exergame in Patients with Metabolic Syndrome

Research Institute, Busan 49241, Korea

16 \* Corresponding author

1

2

3

12

13

- 17 Kyoung-Im Cho, MD, Division of Cardiology, Department of Internal Medicine, Kosin
- University School of Medicine, 34 Amnam-Dong, Seo-Ku, Busan 49267, Korea, Tel: (82) 51-
- 19 990-6105, Fax: (82) 51-990-3005, E-mail: kyoungim74@gmail.com

- 20 \* Co-corresponding author
- 21 **Bo Hyun Kim, M.D., Ph.D.** Department of Internal Medicine, Biomedical Research Institute,
- 22 Pusan National University Hospital, Busan, 49241, Korea. Tel: (82)-51-240-7678, Fax: (82)
- 23 51-254-3237, E-mail: pons71@hanmail.net

24

25

- Abstract
- 27 **Background**: Recent studies indicate that exercise-related games can improve executive
- 28 function, attention processing, and visuospatial skills.
- 29 **Objective:** This study investigates whether exercise with exergaming can improve the
- 30 executive function in patients with metabolic syndrome (MetS).
- 31 **Methods:** Twenty-two MetS patients were recruited and randomly assigned to the exergaming
- 32 group (EXG) and treadmill exercise group (TEG). The reaction time (RT) and
- electrophysiological signal from the frontal (Fz), central (Cz), and parietal (Pz) cortex were
- 34 collected during a Stroop task after 12 weeks' exercise.
- 35 Results: During the Stroop congruence (facilitation) judgment task, both EXG and TEG
- showed significantly faster RT after 12 weeks of exercise training. For N200 amplitude, EXG
- 37 significantly increased on Fz and Cz. These changes were significantly larger in EXG than
- 38 TEG. For P300 amplitude, EXG significantly increased on Fz, Cz, and Pz, while TEG
- 39 significantly increased on Cz and Pz only. During the Stroop incongruence (interference)
- 40 judgment task, both EXG and TEG showed significantly faster RT. For P300 amplitude, EXG

| 41 | significantly increased on Fz and Cz only, while TEG significantly increased on Fz, Cz, and |
|---|---|
| 42 | Pz. |
| 43 | Conclusions: Exergaming improves executive function in patients with MetS as much as |
| 44 | normal aerobic exercise. Particularly, the unique benefit of the exergaming beyond increased |
| 45 | aerobic capacity is the improvement of selective attention among cognitive functions. Thus, |
| 46 | exergaming could be recommended to someone who needs to improve brain responses of |
| 47 | concentration and judgment as well as physical fitness. |
| 48 | <b>Keywords</b> : exergaming; executive functions; event-related potential; metabolic syndrome |
| 49 | |
| 50 | |
| 51 | |
| 52 | |
| 53 | |
| 54 | |
| 55 | |
| 56 | |
| 57 | |
| 58 | |
| 59 | |
| 60 | |

#### Introduction

61

62

63

64

65

66

67

68

69

70

71

72

73

74

75

76

77

78

79

80

81

82

83

In recent years, the relationship between cognitive function and metabolic syndrome has been widely studied [1,2]. Metabolic syndrome (MetS) has been shown to be associated with a decline in executive function [3,4] due to multiple risk factors, including hypertension, dyslipidemia, impaired glucose homeostasis, and abdominal obesity. Executive functions include basic cognitive processes such as attentional control, cognitive inhibition, inhibitory control, working memory, and cognitive flexibility [5]. Cognitive neuroscience is using Stroop tasks to measure selective attention capacity and skills, as well as processing speed ability, indicating executive functions [6]. Electroencephalographic (EEG) activity using event-related positioning technology P300 and N200 has been widely used to measure selective attention capacity and skills, and a behavioral performance such as reaction time (RT) is commonly used to measure processing speed ability [7,8]. N200 negativity (200~350 ms post-stimulus) is an event-related potential (ERP), which indicates attentional capacity that is usually induced before motion response control and is related to the cognitive processes of stimulus recognition and differentiation [9]. P300 positivity (300~600 ms post-stimulus) is another ERP, reflecting memory-related neural processing that is involved in categorizing incoming information and updating the context of the working memory (e.g., encoding, rehearsal, recognition, and retrieval) [10]. It is well known that aerobic exercise training provides various beneficial clinical outcomes in metabolic disease patients [11,12]. Its effects on cognitive function, especially executive function, also have been reported [13]. Furthermore, recent studies reported that both aerobic and resistance exercise training facilitate overall electrophysiological effects (e.g., increased ERP P300 amplitudes) and behavior index (e.g., faster RT) in healthy elderly people [14,15].

In addition, aerobic exercise has also been reported to improve cognitive processes in cortical cognitive control (P300 amplitude) in studies of chronic stroke patients [16].

Recently, exergaming (a combination of "exercise" and "gaming") has attracted much attention as a novel exercise method to improve cognitive function because it utilizes video games that require body movements while simultaneously presenting the user with a cognitively challenging environment [17]. Along with its popular usage for leisure and entertainment, there is a growing interest in the application of exergaming to improve clinical outcomes. Recent studies using exergaming showed beneficial effects on cognitive and dual-task functions, which reduced falls in older adults [18] as well as cardiovascular disease risks such as body fat, serum adipokine levels, and lipid profiles [19]. Exergaming also promoted executive functions and cognitive processing speed in elderly and children [20,21]. This growing evidence suggests that exergaming's have the benefit of improving cognitive and physical functions.

Although many previous studies have reported improvements in cognitive function following exergaming, it is not clear whether this benefit is due to an exercise effect or video game effect. In addition, all of these studies measured RT, instead of ERP using EEG, which limits to illuminate brain activities. Considering that EEG can measure electrical activities in various cortex areas in the brain, it is necessary to investigate ERP using EEG to evaluate executive function. Therefore, we examined the benefits of exergaming compared to normal exercise and investigated executive function by measuring RT as well as N200 and P300 in three cortex areas during Stroop tasks in patients with MetS.

#### Methods

106

107

108

109

110

111

112

113

114

115

116

117

118

119

120

125

#### **Participants**

A total of 22 MetS male and female patients aged between 50-80 years participated in this study. MetS was defined according to the modified NCEP Adult Treatment Panel III (NCEP-ATP III) definition for South Asians. Briefly, individuals with three or more of the following criteria were defined as MetS: central obesity (waist circumference ≥90 cm for men; ≥ 85 cm for women), fasting plasma glucose ≥100 mg/dL or current treatment for diabetes mellitus, systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg or current treatment for hypertension, serum triglyceride ≥150 mg/dL, low HDL cholesterol (men<40 mg/dL; women<50 mg/dL) [22]. Subjects were asked to not exercise for 24 hours before the experiment. They were also instructed to eat usual meals and to finish meals 4 hours before the experiment, while avoiding alcohol 1 day before the experiment and caffeine during the 4 hours prior to the experiment. All subjects were required to complete a written informed consent approved by the Institutional Review Board of Kosin University College of Medicine.

- The sample size was calculated using sample size calculation software (G\*Power version
- 3.1.9.2 for Windows; <a href="http://www.gpower.hhu.de">http://www.gpower.hhu.de</a>), with effect size 0.484, statistical power 0.8,
- and statistical level of significance 0.05. This effect size was calculated from the previous
- studies [13,14]. As a result, the sample size for each group became 8, and we decided to recruit
- 124 11 patients for each group, with a potential 30% dropout rate.

#### **Exercise Training Interventions**

- Exercise training was conducted at the Kosin University Gospel Hospital U-healthcare Center.
- Each participant was instructed to immediately inform the supervisor if he or she experienced
- any unusual symptoms during exercise training and to consult a physician if needed. Subjects

were excluded if they did not perform more than 80% of the exercise sessions.

All subjects were randomly divided into two groups: exergaming and treadmill exercise group. Subjects had 2 weeks of adaptation and then carried out 12 weeks of exercise training: 60 min/day, 60-80% of heart rate reserved (HRR), 3 days/week. Each exercise session consisted of 10 minutes of warm-up, 40 minutes of main exercise, and 10 minutes of warm-down. The exergaming group (EXG) performed exercise using Exerheart® devices (D&J Humancare, Busan, South Korea) composed of a running/jumping mat  $[730(W) \times 730(D) \times 130(H)]$  and a tablet PC on a stand (can be adjusted to any height between 70 and 155 cm) (Supplemental Figure 1A). Exerheart® is an exergaming developed for in-situ running along with the video game called "Alchemist's Treasure" (D&J Humancare, Busan, South Korea) (Supplemental Figure 1B). To play this game, the subject has to run or jump on a spot on the mat to move a virtual avatar on the screen of the tablet PC to the front, back, left, and right along with music (Supplemental Video 1 for online). The subject can control the speed of avatar movement by running or jumping speed on the mat. The treadmill exercise group (TEG) performed exercise using commercial treadmills (MOTUS, Gyeonggi-do, South Korea). Each subject walked or ran on the treadmill at a comfortable speed. For both EXG and TEG, all subjects' heart rates (HR) during exercise were monitored using HR monitors (polar RS400sd, Madison Height, Michigan, USA) to confirm that the value was within the target HR range. The Karvonen formula (1957) [23] was used to calculate HR reserve (HRR, estimated maximal HR- resting HR) and target HR during exercise [(HRR ×

#### **Stroop Test**

129

130

131

132

133

134

135

136

137

138

139

140

141

142

143

144

145

146

147

148

149

150

given percentage of training intensity) + resting HR)].

For assessment of executive function, a computer-based version of the Stroop task was administered with Telescan software (LAXTHA, Daejeon, South Korea). During the task, subjects were presented with a color word appearing in the same color on congruent trials (e.g. "blue" printed in blue) and in a different color on incongruent trials (e.g. "blue" printed in green) [24]. To provide similar visual content, blue, green, and yellow were chosen as stimuli.

Subjects performed Stroop task twice, pre- and post-exercise training. Subjects sat 1 meter from the screen, and when the color words appeared on the screen, they clicked the left keyboard for the congruent test and the right keyboard for the incongruent test. Subjects were instructed to respond as quickly and accurately as possible. The rate of measurement targeted for 50%. Each color word (vertical viewing angle: 2 °) was presented for 200 ms, and the

response was allowed within 1500 ms. The inter-stimulus interval varied randomly between

### **Electroencephalographic (EEG) Measurements**

1500 and 2500 ms.

EEG activity was recorded during the modified Stroop task using a computerized polygraph system— Type A: A total of 31-channel Poly G-A (LAXTHA, Daejeon, South Korea). Ag-AgCl electrodes (LAXTHA, Daejeon, South Korea) were placed on frontal (Fz), central (Cz), and parietal (Pz) cortex areas, according to the International 10-20 system. Midline locations referenced to link earlobe electrodes. Horizontal and vertical electrooculograms (EOGs) were monitored by electrodes placed above and below the left eye and at the outer canthus of both eyes, respectively. The impedance of all electrodes was maintained below  $10 \, k\Omega$ . The bandpass filter of the amplifier was 0.1– $100 \, Hz$ , the sampling rate was  $1000 \, Hz$ , and a notch filter was at  $60 \, Hz$ .

The N200 component was defined as the largest positive peak occurring between 200-350 ms

post-stimulus, and the P300 component was defined as the largest positive peak occurring between 300~600 ms post-stimulus [7]. N200 and P300 amplitudes were measured as the difference between the mean pre-stimulus baseline and maximum peak amplitude. Telescan's built-in high pass IIR filter was used for filtering. Waveforms were digitally smoothed with a low-pass filter using a half-power cut-off of 10 Hz prior to analysis.

#### **Statistical Analysis**

Due to the small sample size, we used nonparametric statistics for data analysis. We used the Wilcoxon signed-rank test to examine the changes of each dependent variable after intervention within each group. The Mann–Whitney U test was used to make comparisons of the delta values between training groups ( $\Delta$ -EXG vs  $\Delta$ -TEG). The effect size of partial eta-squared ( $\eta$ 2) was reported for significant effects, where the alpha level for all of the tests was set at 0.05. Data were expressed as mean  $\pm$  standard deviation of mean. All statistical tests were processed using the software SPSS 24 version.

#### **Results**

Demographic and physical characteristics for all subjects are provided in Table 1. There were no significant group differences at baseline measurements.

#### Reaction Time

The changes in congruent RT after 12 weeks of exercise training were not significantly different between EXG and TEG (Table 2). EXG significantly shortened congruent RT, as did TEG (Figure 1A). The changes in incongruent RT after 12 weeks of exercise training were not significantly different between EXG and TEG. EXG significantly shortened incongruent RT, as did TEG (Figure 1B).

## Event-related Potential Data

197

198 N200 amplitude The results in Table 3 after 12 weeks of exercise training, the increases in congruent N200 199 amplitude on Cz, and Pz in EXG were significantly greater than in TEG, but not on Fz. EXG 200 significantly increased congruent N200 amplitude on Cz, but not on Fz and Pz. On the other 201 hand, TEG showed no significant changes in congruent N200 amplitude on Fz, Cz, or Pz 202 203 (Figure 2A). The changes in incongruent N200 amplitude on Fz, Cz, and Pz after 12 weeks of exercise 204 training were not significantly different between EXG and TEG (Table 3). Interestingly, EXG 205 did not significantly change incongruent N200 amplitude on Fz, Cz, or Pz. TEG also did not 206 significantly change incongruent N200 amplitude on Fz, Cz, or Pz (Figure 2B). The waveforms 207 208 of congruent and incongruent N200 amplitudes on Fz, Cz, and Pz for EXG and TEG before and after exercise are shown in Figure 3. 209 P300 amplitude 210 211 Table 3 shows the results of Mann-Whitney U test for changes in congruent P300 amplitude on Fz, Cz, and Pz after 12 weeks of exercise training was not significantly different between 212 213 EXG and TEG. EXG significantly increased congruent P300 amplitude on Fz, Cz, and Pz. However, TEG significantly increased congruent P300 amplitude on only Fz and Cz, but not 214 on Pz (Figure 2C). 215 There were no significant differences in the changes in incongruent P300 amplitude on Fz, Cz, 216 and Pz between EXG and TEG after 12 weeks of exercise training (Table 3). EXG significantly 217 increased incongruent P300 amplitude on Cz and Pz, but not on Fz. On the other hand, TEG 218

significantly increased incongruent P300 amplitude on Fz, Cz, and Pz (Figure 2D). The waveforms of congruent and incongruent P300 amplitudes on Fz, Cz, and Pz for EXG and TEG before and after exercise are shown in Figure 3.

#### Discussion

219

220

221

222

223

224

225

226

227

228

229

230

231

232

233

234

235

236

237

238

239

240

241

This study was the first to investigate the benefits of exergaming compared to normal exercise on the behavioral performance and executive function of patients with MetS. We found that 12 weeks of both exergaming and treadmill exercise training similarly and effectively improved behavioral performance and congruent and incongruent memory-related neural processing. However, only exergaming training improved congruent selective attention, while neither exergaming nor treadmill exercise training affected incongruent selective attention. These results suggest similar overall effects of exergaming and normal exercise on behavioral performance and executive function of patients with MetS, but exergaming could be more effective than normal exercise for congruent selective attention. The present study showed that both 12 weeks of exergaming and treadmill exercise training effectively improved reaction time in MetS patients, and these changes were not different between exergaming and treadmill exercise training. These results indicate that both exergaming and normal exercise improve behavioral performance, but exergaming does not have more beneficial effects compared to normal exercise. In our previous study, we examined the performance of control tasks using a simple acute aerobic exercise and complex exercise [25]. The results indicated that participants did not have different performance when participating in simple exercise compared to very skilled complex exercises. In another study, contrary to our results, an acute single-bout study comparing the effects of standard normal exercise to exergaming on attention performance in young adults found no significant

improvement with exergaming [7]. The result of that study suggests that, after 20 minutes of unskilled Wii Fit TM, the brain needs more information processing, which may be the source of control requirements and pressure increases, offsetting the potential benefits of the exercise component. However, compared to the Wii Fit<sup>TM</sup>, exergaming with exerheart® is runningbased aerobic exercise on an air cushion board with game-based contents such as adventures, racing, and quizzes, which continue to arouse interest in exercise. So, with exerheart®, an individual is running constantly with changing visual stimuli; these repeated effects will simultaneously increase physical activity and cognitive function via interactive virtual reality engagement [20]. Therefore, through exergaming and treadmill exercise, the reaction time of Stroop task conditions of MetS patients could be shortened, which would promote basic information processing and executive function of suppression control. In this study, the congruent and incongruent P300 amplitudes were increased after both 12 weeks of exergaming and treadmill exercise training, with no difference between EXG and TEG. These results indicate that both exergaming and normal exercise improve memoryrelated neural processing, but exergaming has no more beneficial effects than normal exercise. In other words, participation in exercise, regardless of exercise modality, induces an increase in working memory in executive function. However, our previous study showed that P300 amplitude increased during a control task following futsal relative to seated rest or treadmill exercise, indicating that complex control of the brain stimulates the executive control network of the cortex [25]. It was found that, as age increases, the P300 amplitude in the central (Cz) region decreases, and the scalp distribution of the P300 amplitude is transferred to the frontal region [26]. Pontifex et al. [27] examined P300 components and found that older adults with

242

243

244

245

246

247

248

249

250

251

252

253

254

255

256

257

258

259

260

261

262

high cardiorespiratory fitness only exhibited greater P300 amplitudes, and Tsai and colleagues [28] found that different exercise types have greater amplitudes for older P300. However, as they pointed out, regardless of the type of older people to participate in sports, physical exercise is a lifestyle factor that is crucial to preventing age-related biological degeneration in the frontal-to-parietal areas, thus delaying the cognitive declines associated with later life. Considering that exergaming is a kind of aerobic exercise, it stands to reason that exergaming could improve not only cardiovascular health, but also cognitive plasticity, thereby improving categorization of incoming information and updating the context of working memory in MetS patients. We found that neither exergaming nor treadmill exercise training affected incongruent N200 amplitude. However, the consistent N200 amplitude only increased by exergaming training. These results indicate that, while neither exergaming nor normal exercise affects incongruent selective attention, only exergaming improves congruent selective attention, which suggests that exergaming have a more beneficial effect on congruent selective attention compared to normal exercise. The results of many studies on the relationship between exercise and N200 amplitude indicate show that exercise has no significant effect on N200 amplitude [28,29]. Pontifex and his colleagues showed that general decreases in N200 amplitudes across scalp sites were observed during exercise relative to rest [29]. The N200 component plays a key role in the anterior cingulate cortex (ACC), which is part of the potential prefrontal cortex and regulates dopaminergic neurons in cognitive functions, such as working memory, attention, and decision making [30-32]. Therefore, the reduction of N200 amplitude caused by normal aerobic exercise severely limits ACC activity [29]. In light of our N200 amplitude findings, these

264

265

266

267

268

269

270

271

272

273

274

275

276

277

278

279

280

281

282

283

284

285

286

results suggest that exergaming better regulates the activity of ACC in the prefrontal cortex

than aerobic exercise, thereby effectively increasing consistent selective attention.

287

288

289

290

291

292

293

294

295

296

297

298

299

300

301

302

303

304

305

306

307

308

309

Recent studies suggest that combining motor and cognitive demands during exercising can improve cognitive function more than training these domains separately [17,33]. In addition, cognitive video game training can have beneficial effects on memory, attention, and reaction time in older adults [34,35]. In previous studies, when participants consistently performed exercises in a virtual environment, an increase in N200 amplitude positively promoted decision-making (frontal and central) and visual perception (occipital) [36]. Therefore, the exergaming positively promotes visual perceptual stimulation in the virtual environment to enhance the selective attention activity associated with the cerebral cortex, thereby strongly promoting executive function. Exercise and video games can each improve brain structure and function [37-40]; thus, their combination can have a complementary effect on brain stimulation and protection. Our study provides evidence that exergaming improves reaction time and incongruent memoryrelated neural processing in MetS patients as much as normal aerobic exercise. In addition, exergaming improves congruent selective attention, which was not changed by normal aerobic exercise. Therefore, exergaming could provide an innovative way to enjoy aerobic exercise compared to repetitive, conventional exercises. Although this study found significant results, there are some limitations in this study as follows:

Although this study found significant results, there are some limitations in this study as follows:

1) the sample size in this study is relatively small, even though all patients were very hard motion for 12 weeks; 2) the range of age was relatively large, 50~80 years old. Considering that with age, response time and brain activity are usually slower, we cannot rule out the possibility that age will affect the performance of executive function. However, the mean age was similar in both groups, so this possibility might be low in this study; 3) the intensity of the

310 Exerheart® using "Alchemist's Treasure" game was not able to be controlled. 311 **Conclusions** 312 The results of this study suggest that exergaming enhances brain response to concentration and 313 judgment, resulting in increased behavioral response of the MetS patients, comparable to that 314 of normal aerobic exercise. Furthermore, the unique advantage of exergaming is that it 315 improves selective attention among cognitive functions, unlike normal aerobic exercise. 316 Therefore, exergaming could be recommended to some patients who need to improve executive 317 function as well as physical fitness. 318 319 Acknowledgments. We thank the participants for their time and effort while participating in 320 the present study. The authors declare that the results of the study are presented clearly, honestly, 321 and without fabrication, falsification, or inappropriate data manipulation. The authors declare 322 that there are no conflicts of interest. 323 324 325 Funding. This research did not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors. 326 327 328 **Conflicts of Interest** None declared. 329

#### Multimedia Appendix 1. MP4.

- Participants played the video game with Exerheart®.
- 333 [Author- Kyoung Im Cho, videographer Shanshan Wu, 15 seconds length and 1.48 MB size]

334

335

331

#### References

- González HM, Tarraf W, Vásquez P, Sanderlin AH, Rosenberg NI, Davis S, et al. Metabolic Syndrome and Neurocognition Among Diverse Middle-Aged and Older Hispanics/Latinos: HCHS/SOL Results. Diabetes Care 2018 Jul;41(7):1501-1509. [doi:10.2337/dc17-1896] [Medline: 29716895]
- Shigaeff N, Amaro E, Franco FGM, Jacinto AF, Chiochetta G, Cendoroglo MS, et al. Functional magnetic resonance imaging response as an early biomarker of cognitive decline in elderly patients with metabolic syndrome. Arch Gerontol Geriatr 2017 Nov;73:1-7.[doi:10.1016/j.archger.2017.07.002] [Medline: 28711765]
- Falkowski J, Atchison T, Debutte-Smith M, Weiner MF, O'Bryant S. Executive functioning and the metabolic syndrome: a project FRONTIER study. Arch Clin Neuropsychol 2014 Feb;29(1):47-53. [doi: 10.1093/arclin/act078] [Medline: 24152591]
- Bokura H, Nagai A, Oguro H, Kobayashi S, Yamaguchi S. The association of metabolic syndrome with executive dysfunction independent of subclinical ischemic brain lesions in Japanese adults. Dement Geriatr Cogn Disord 2010;30(6):479-85. [doi: 10.1159/000322057] [Medline: 21252541]
- Royall DR, Lauterbach EC, Cummings JL, Reeve A, Rummans TA, Kaufer DI, et al. Executive control function: a review of its promise and challenges for clinical research. A report from the Committee on Research of the American Neuropsychiatric Association. J Neuropsychiatry Clin Neurosci 2002 Fall;14(4):377-405. [DOI: 10.1176/jnp.14.4.377] [Medline: 12426407]
- Badzakova-Trajkov G, Barnett KJ, Waldie KE, Kirk IJ. An ERP investigation of the Stroop task: the role of the cingulate in attentional allocation and conflict resolution.
  Brain Res 2009 Feb 9;1253:139-48. [doi: 10.1016/j.brainres.2008.11.069] [Medline: 19084509]
- Patel SH, Azzam PN. Characterization of N200 and P300: selected studies of the Event-Related Potential. Int J Med Sci 2005;2(4):147-54. [Medline: 16239953]
- Thorpe S, Fize D, Marlot C. Speed of processing in the human visual system. Nature 1996 Jun 6;381(6582):520-2. [doi:10.1038/381520a0] [Medline: 8632824]
- Dennis TA, Chen CC. Neurophysiological mechanisms in the emotional modulation of attention: the interplay between threat sensitivity and attentional control. Biol Psychol 2007 Sep;76(1-2):1-10. [doi:10.1016/j.biopsycho.2007.05.001] [Medline: 17582673]
- 367 10 Polich J. Updating P300: an integrative theory of P3a and P3b. Clin Neurophysiol 2007 368 Oct;118(10):2128-48. [doi:10.1016/j.clinph.2007.04.019] [Medline: 17573239]
- Wewege MA, Thom JM, Rye KA, Parmenter BJ. Aerobic, resistance or combined

- training: A systematic review and meta-analysis of exercise to reduce cardiovascular risk in adults with metabolic syndrome. Atherosclerosis 2018 Jul;274:162-171. [doi:10.1016/j.atherosclerosis.2018.05.002] [Medline: 29783064]
- Lemes IR, Turi-Lynch BC, Cavero-Redondo I, Linares SN, Monteiro HL. Aerobic training reduces blood pressure and waist circumference and increases HDL-c in metabolic syndrome: a systematic review and meta-analysis of randomized controlled trials. J Am Soc Hypertens 2018 Aug;12(8):580-588. [doi:10.1016/j.jash.2018.06.007] [Medline: 29945775]
- Fong DY, Chi LK, Li F, Chang YK. The benefits of endurance exercise and Tai Chi Chuan for the task-switching aspect of executive function in older adults: an ERP study. Front Aging Neurosci 2014 Oct 28;6:295. [doi:10.3389/fnagi.2014.00295] [Medline: 25389403]
- Tsai CL, Pan CY, Chen FC, Tseng YT. Open- and Closed-Skill Exercise Interventions Produce Different Neurocognitive Effects on Executive Functions in the Elderly: A 6-Month Randomized, Controlled Trial. Front Aging Neurosci 2017 Sep 12;9:294. [doi:10.3389/fnagi.2017.00294] [Medline: 28959200]
- Tsai CL, Wang WL. Exercise-mode-related changes in task-switching performance in the elderly. Front Behav Neurosci 2015 Mar 6;9:56. [doi:10.3389/fnbeh.2015.00056] [Medline: 25798097]
- Swatridge K, Regan K, Staines WR, Roy E, Middleton LE. The Acute Effects of Aerobic Exercise on Cognitive Control among People with Chronic Stroke. J Stroke Cerebrovasc Dis 2017 Dec;26(12):2742-2748. [doi:10.1016/j.jstrokecerebrovasdis.2017.06.050] [Medline: 28774794]
- Limperos AM, Schmierbach M. Understanding the Relationship Between Exergame Play Experiences, Enjoyment, and Intentions for Continued Play. Games Health J 2016 Apr;5(2):100-7. [doi:10.1089/g4h.2015.0042] [Medline: 26871873]
- Fu AS, Gao KL, Tung AK, Tsang WW, Kwan MM. Effectiveness of Exergaming Training in Reducing Risk and Incidence of Falls in Frail Older Adults With a History of Falls. Arch Phys Med Rehabil. 2015 Dec;96(12):2096-102. [doi: 10.1016/j.apmr.2015.08.427] [Medline: 26360975]
- 400 19 Amorim MGS, de Oliveira MD, Soares DS, da Silva Borges L, Dermargos A, Hatanaka E. Effects of exergaming on cardiovascular risk factors and adipokine levels in women.

  J Physiol Sci 2018 Sep;68(5):679. [doi:10.1007/s12576-017-0581-5] [Medline: 29305789]
- Dimitrova J, Hogan M, Khader P, O'Hora D, Kilmartin L, Walsh JC, et al. Comparing the effects of an acute bout of physical exercise with an acute bout of interactive mental and physical exercise on electrophysiology and executive functioning in younger and older adults. Aging Clin Exp Res 2017 Oct;29(5):959-967. [doi:10.1007/s40520-016-0683-6] [Medline: 27866346]
- Benzing V, Schmidt M. Cognitively and physically demanding exergaming to improve executive functions of children with attention deficit hyperactivity disorder: a randomised clinical trial. BMC Pediatr 2017 Jan 10;17(1):8. [doi:10.1186/s12887-016-0757-9] [Medline: 28068954]
- Pandit K, Goswami S, Ghosh S, Mukhopadhyay P, Chowdhury S. Metabolic syndrome in South Asians. Indian J Endocrinol Metab 2012 Jan-Feb;16(1):44–55 [doi:10.4103/2230-8210.91187] [Medline: 22276252]
- Karvonen MJ, Kentala E, Mustala O. The effects of training on heart rate; a longitudinal

- 417 study. Ann Med Exp Biol Fenn 1957;35(3):307-15. [Medline: 13470504]
- Ilan AB, Polich J. P300 and response time from a manual Stroop task. Clin Neurophysiol 1999 Feb;110(2):367-73. [Medline: 10210626]
- Won J, Wu SS, Ji HQ, Smith JC, Park J. Executive Function and the P300 after Treadmill Exercise and Futsal in College Soccer Players. Sports (Basel) 2017 Sep 26;5(4). [doi:10.3390/sports5040073] [Medline: 29910433]
- Picton TW, Stuss DT, Champagne SC, Nelson RF. The effects of age on human eventrelated potentials. Psychophysiology 1984 May;21(3):312-25. [Medline: 6739673]
- Pontifex MB, Hillman CH, Polich J. Age, physical fitness, and attention: P3a and P3b. Psychophysiology 2009 Mar;46(2):379-87. [doi:10.1111/j.1469-8986.2008.00782.x] [Medline: 19170947]
- Tsaia CL, Wang CH, Pan CY, Chen FC, Huang SY, Tseng YT. The effects of different exercise types on visuospatial attention in the elderly. Psychol Sport Exerc 2016 Sep; 26, 130-138, [doi:10.1016/j.psychsport.2016.06.013]
- Pontifex MB, Hillman CH. Neuroelectric and behavioral indices of interference control during acute cycling. Clin Neurophysiol 2007 Mar;118(3):570-80. [doi:10.1016/j.clinph.2006.09.029] [Medline: 17095295]
- Buzzell GA, Fedota JR, Roberts DM, McDonald CG. The N2 ERP component as an index of impaired cognitive control in smokers. Neurosci Lett 2014 Mar 20;563:61-5. [doi:10.1016/j.neulet.2014.01.030] [Medline: 24486891]
- Seamans JK, Yang CR. The principal features and mechanisms of dopamine modulation in the prefrontal cortex. Prog Neurobiol 2004 Sep;74(1):1-58. [doi:10.1016/j.pneurobio.2004.05.006] [Medline: 15381316]
- Tritsch NX, Sabatini BL. Dopaminergic modulation of synaptic transmission in cortex and striatum. Neuron 2012 Oct 4;76(1):33-50. [doi:10.1016/j.neuron.2012.09.023] [Medline: 23040805]
- Fabre C, Chamari K, Mucci P, Masse-Biron J, Prefaut C. Improvement of cognitive function by mental and/or individualized aerobic training in healthy elderly subjects.

  Int J Sports Med 2002 Aug;23(6):415-21. [doi:10.1055/s-2002-33735] [Medline: 12215960]
- Lauenroth A, Ioannidis AE, Teichmann B. Influence of combined physical and cognitive training on cognition: a systematic review. BMC Geriatr 2016 Jul 18;16:141. [doi:10.1186/s12877-016-0315-1] [Medline: 27431673]
- Oswald WD, Gunzelmann T, Rupprecht R, Hagen B. Differential effects of single versus combined cognitive and physical training with older adults: the SimA study in a 5-year perspective. Eur J Ageing 2006 Nov 10;3(4):179. [doi:10.1007/s10433-006-0035-z] [Medline: 28794762]
- Vogt T, Herpers R, Scherfgen D, Struder HK, Schneider S. Neuroelectric adaptations to cognitive processing in virtual environments: an exercise-related approach. Exp Brain Res 2015 Apr;233(4):1321-9. [doi:10.1007/s00221-015-4208-x] [Medline: 25630906]
- Deslandes A, Moraes H, Ferreira C, Veiga H, Silveira H, Mouta R, et al. Exercise and mental health: many reasons to move. Neuropsychobiology 2009;59(4):191-8. [doi:10.1159/000223730] [Medline: 19521110]
- Shams TA, Foussias G, Zawadzki JA, Marshe VS, Siddiqui I, Müller DJ, et al. The Effects of Video Games on Cognition and Brain Structure: Potential Implications for Neuropsychiatric Disorders. Curr Psychiatry Rep 2015 Sep;17(9):71. [doi:10.1007/s11920-015-0609-6] [Medline: 26216589]

| 464<br>465 | 39 | Wang P, Zhu XT, Qi Z, Huang S, Li HJ. Neural Basis of Enhanced Executive Function in Older Video Game Players: An fMRI Study. Front Aging Neurosci 2017 Nov |
|---|---|---|
| 466<br>467 | 40 | 21;9:382. [doi:10.3389/fnagi.2017.00382] [Medline: 29209202] Zhang X, Ni X, Chen P. Study about the effects of different fitness sports on cognitive |
| 468 | 10 | function and emotion of the aged. Cell Biochem Biophys 2014 Dec;70(3):1591-6. |
| 469<br>470 | | [doi:10.1007/s12013-014-0100-8] [Medline: 24997050] |
| 170 | | |
| 471 | | |
| 472 | | |
| 473 | | |
| 474 | | |
| 47E | | |
| 475 | | |
| 476 | | |
| 477 | | |
| 478 | | |
| 479 | | |
| 480 | | |
| .00 | | |
| 481 | | |
| 482 | | |
| 400 | | |
| 483 | | |
| 484 | | |
| 485 | | |
| . 55 | | |

## Figure 1. Mean reaction time (RT) during stroop task (A. congruent/ B. incongruent) 487 performance after exergaming group (EXG) and treadmill exercise group (TEG) before and 488 after the exercise intervention. 489 Figure 2. N200 and P300 amplitudes (mean $\pm$ SE) on three electrodes (Fz, Cz, and Pz) during 490 the Stroop task (A. congruent/B. incongruent N200 amplitudes; C. congruent/D. incongruent 491 P300 amplitudes) in the exergaming group (EXG) and treadmill exercise group (TEG) before 492 and after 12 weeks of exercise training. 493 494 495 Figure 3. Average event-related potential waveforms of electrodes (Fz, Cz, Pz) for mean N200 and P300 amplitudes during the Stroop test (A. congruent/ B. incongruent) in the exergaming 496 group (EXG) and treadmill exercise group (TEG) before and after 12 weeks of the exercise 497 training. 498 499 500 Supplement Figure 1. A. The exergaming group performed exercise using Exerheart® devices by permission of D&J Humancare which had the copyright holder of Exerheart®. B. Features 501 of the video game "Alchemist's Treasure". 502 503 504 505

**Figure Legends** 

486

Table 1. Baseline characteristics of demographic information.

| Group | EXG (N=11) | TEG(N=11) | P value |
|-------------------|--------------------|--------------------|---------|
| Factor | EAU (N-11) | 1EG(N-11) | r value |
| Age(years) | 64±10 | $60 \pm 7$ | .298 |
| Height(cm) | 154.24±5.73 | 161.66±7.1 | .014 |
| Weight(kg) | 69.38±10.54 | 71.47±11.62 | .663 |
| $BMI(kg/m^2)$ | 29.07±3.3 | $27.31\pm3.52$ | .24 |
| WC(cm) | 97.36±10.95 | 93.6±8.78 | .399 |
| Glucose(mg/dl) | 123.55±25.68 | 112.36±29.37 | .353 |
| HDL-chol (mmol/L) | 46.32±8.91 | $50.59 \pm 10.52$ | .316 |
| LDL-chol (mmol/L) | 66.19±22.8 | $78.38 \pm 19.52$ | .193 |
| TC (mmol/L) | 134.81±25.52 | $146.67 \pm 12.04$ | .179 |
| TG (mmol/L) | 136.82±78.88 | 145.73±142.74 | .858 |
| SBP (mmHg) | $127.09 \pm 16.86$ | 128.09±17.39 | .892 |
| DBP (mmHg) | 75.55±9.43 | 77.73±11.99 | .64 |

Values are mean  $\pm$  SD. EXG, exergame group; TEG, treadmill exercise group; BMI, body mass index; WC, waist circumference; TG, triglycerides; HDL-chol, high-density lipoprotein cholesterol; LDL-chol, low-density lipoprotein cholesterol; SBP, systolic blood pressure; DBP, diastolic blood pressure.

# Table 2. Comparison of Stroop task congruent and incongruent reaction time of EXG and TEG groups

| Effects | Group | pre | post | P value <sup>a</sup> | η2 | P value <sup>b</sup> |
|---|---|---|---|---|---|---|
| Congruent | EXG | 1265.91±383.15 | 1012.09±221.64 | 0.003 | 0.053 | 0.279 |
| Congruent | TEG | 1124.18±161.21 | 957.82±138.05 | 0.003 | 0.033 | |
| Incongruent | EXG | 1299.09±367.48 | 984.73±204.81 | 0.003 | 0.008 | 0.670 |
| Incongruent | TEG | 1171.36±163.26 | 974.55±120.97 | 0.003 | U.U08 | |

<sup>&</sup>lt;sup>a</sup> Wilcoxon Signed Rank Test: comparison pre vs. post within group.

<sup>&</sup>lt;sup>b</sup> Mann Whitney U Test: comparison the delta values between groups (Δ-EXG vs Δ-TEG).

Table 3. Comparison of Stroop task congruent and incongruent N200 / P300 amplitudes of EXG and TEG groups

| Components | Effects | | Group | pre | post | P value <sup>a</sup> | η2 | P value <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|
| | Congruent | Fz | EXG | -1.33±1.95 | -4.1±3.02 | 0.091 | 0.138 | 0.088 |
| | | | TEG | -0.98±3.14 | -0.41±3.82 | 0.328 | | |
| | | Cz | EXG | -1.59±2.54 | -5.13±2.94 | <mark>0.016</mark> | 0.291 | 0.010 |
| | | CZ | TEG | -1.61±3.89 | -0.97±4.59 | 0.424 | | |
| | | Pz | EXG | -1.58±1.89 | -4.06±2.89 | 0.062 | 0.207 | 0.034 |
| N200 | | | TEG | -1.32±3.62 | -0.89±3.99 | 0.534 | | |
| Amplitude | 2 | Fz | EXG | -2.85±2.3 | -2.78±3.02 | 0.477 | 0.041 | 0.365 |
| | | | TEG | -1.37±3.3 | -0.73±3.18 | 0.424 | | |
| | Inconomicant | | EXG | -3.23±2.69 | -3.93±2.92 | 0.286 | 0.099 | 0.151 |
| | Incongruent | Cz | TEG | -1.9±3.82 | -1.1±3.65 | 0.213 | | |
| | | Pz | EXG | -2.86±2.45 | -3.07±2.62 | 0.722 | 0.008 | 0.699 |
| | | | TEG | -1.4±3.66 | -1.01±3.52 | 0.477 | | |
| | Congruent | Fz | EXG | 2.3±1.94 | 7.12±5.73 | 0.003 | 0.008 | 0.699 |
| | | | TEG | 3.21±1.95 | $4.82\pm3.78$ | 0.011 | | |
| | | Cz | EXG | 1.92±1.63 | 6.49±5.28 | 0.004 | 0.006 | 0.748 |
| | | | TEG | $2.36\pm0.93$ | $5.08 \pm 3.03$ | 0.013 | | |
| | | Pz | EXG | 1.44±1.69 | 5.2±5.88 | 0.004 | 0.099 | 0.151 |
| P300 | | | TEG | 1.74±1.26 | $4.87 \pm 3.64$ | 0.328 | | |
| amplitude | Incongruent | Fz | EXG | 2.26±3.14 | 4.48±3.27 | 0.091 | 0.018 | 0.562 |
| | | | TEG | 1.93±2.26 | $3.85\pm3.04$ | 0.004 | | |
| | | Cz | EXG | 2.03±2.8 | 4.38±2.81 | <mark>0.016</mark> | 0.002 | 0.847 |
| | | | TEG | 1.59±1.63 | $3.74\pm2.99$ | 0.021 | | |
| | | D- | EXG | 1.58±2.44 | 3.2±2.73 | 0.021 | 0.000 | 0.040 |
| | | Pz | TEG | 1.05±0.92 | $3.33\pm2.59$ | 0.033 | | 0.949 |

<sup>&</sup>lt;sup>a</sup> Wilcoxon Signed Rank Test: comparison pre vs. post within group.
<sup>b</sup> Mann Whitney U Test: comparison the delta values between groups (Δ-EXG vs Δ-TEG).